CLINICAL TRIAL: NCT01042574
Title: The Efficacy and Safety of Cleviprex in Ventriculostomy Patients Requiring IV Antihypertensive Therapy Investigator Initiated Trial
Brief Title: The Efficacy and Safety of Cleviprex in Ventriculostomy Patients Requiring IV Antihypertensive Therapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to secure funding
Sponsor: Methodist Healthcare (Other)
Collaborators: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cleviprex Use In ICB Patients
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2018-03

CONDITIONS: Hypertension; Intracranial Hemorrhage; Subarachnoid Hemorrhage
Keywords: intracranial hemorrhage (ICH); subarachnoid hemorrhage (SAH); intracranial monitoring; external ventricular drain (ventriculostomy); hypertension
MeSH Terms: conditions — Hypertension; Intracranial Hemorrhages; Subarachnoid Hemorrhage | interventions — clevidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Clevidipine butyrate — Cleviprex will be administered according to current package insert instructions, with a starting dose of 2.0mg/hr for 1.5 minutes and thereafter titrated to lower blood pressure to a target goal of 110 mmHG to 140mmHG.
  Other Names: Cleviprex

SUMMARY:
This study is a single-arm, open label protocol evaluating the use of Cleviprex to rapidly control hypertension in patients who present with intracerebral hemorrhage (ICH) or subarachnoid hemorrhage (SAH), and that require ICP monitoring via ventriculostomy (External Ventricular Drain or EVD).

DETAILED DESCRIPTION:
Inclusion Criteria:

The study population will be comprised of men and non-pregnant women age 18 years or older presenting with ICH or SAH that require ICP monitoring via ventriculostomy, and that require IV antihypertensive therapy to a) reduce the risk re-bleeding in SAH and b) reduce the risk of hematoma expansion over time due to further bleeding.

This study population will require rapid and sustained tight control of blood pressure between 110 to 140 mmHg.

Subjects may be included in the study if they meet all of the following criteria:

1. Age 18 years or older
2. Patient presentation with ICH or SAH, and that require ICP monitoring via ventriculostomy drain.
3. Baseline systolic blood pressure (immediately prior to initiation of Cleviprex) >160 mmHg measured
4. Requires IV antihypertensive therapy to achieve SBP 110 - 140 mmHg
5. Patients with a life expectancy of > 5 hours.
6. Written informed consent from the patient or their legal representative before initiation of any study specific procedures

Exclusion Criteria:

Subjects will be excluded from the study if any of the following exclusion criteria apply prior to enrollment:

1. Receipt of an oral antihypertensive within 2 hours prior to initiation of Cleviprex
2. Receipt of IV nicardipine
3. Glasgow coma score (GCS) of <5 and fixed dilated pupils
4. Expectation that the patient will not tolerate or require > 5 hours of concurrent Cleviprex treatment and ICP monitoring
5. Known or suspected aortic dissection
6. Acute myocardial infarction (AMI) on presentation
7. Positive pregnancy test , known pregnancy or nursing mother
8. Intolerance or allergy to calcium channel blockers
9. Allergy to soybean oil or egg lecithin
10. Known liver failure, cirrhosis or pancreatitis
11. Defective lipid metabolism
12. Severe aortic stenosis
13. Prior directives against advanced life support
14. Participation in other clinical research studies involving the evaluation of investigational drugs or devices within 30 days of enrollment

Patients excluded for any of the above reasons may be re-screened for participation at any time if the exclusion characteristic has changed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Patient presentation with ICH or SAH, and that require ICP monitoring via ventriculostomy drain.
3. Baseline systolic blood pressure (immediately prior to initiation of Cleviprex) >160 mmHg measured
4. Requires IV antihypertensive therapy to achieve SBP 110 to 140 mmHg
5. Patients with a life expectancy of > 5 hours.
6. Written informed consent from the patient or their legal representative before initiation of any study specific procedures

Exclusion Criteria:

1. Receipt of an oral antihypertensive within 2 hours prior to initiation of Cleviprex
2. Receipt of IV nicardipine
3. Glasgow coma score (GCS) of <5 and fixed dilated pupils
4. Expectation that the patient will not tolerate or require > 5 hours of concurrent Cleviprex treatment and ICP monitoring
5. Known or suspected aortic dissection
6. Acute myocardial infarction (AMI) on presentation
7. Positive pregnancy test , known pregnancy or nursing mother
8. Intolerance or allergy to calcium channel blockers
9. Allergy to soybean oil or egg lecithin
10. Known liver failure, cirrhosis or pancreatitis
11. Defective lipid metabolism
12. Severe aortic stenosis
13. Prior directives against advanced life support
14. Participation in other clinical research studies involving the evaluation of investigational drugs or devices within 30 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12-31 (Estimated); Study Completion 2010-12-31 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this trial is the time to achieve the pre-specified SBP target range (110-140) within 30 minutes of the initiation of Cleviprex infusion. | 30 minutes

SECONDARY OUTCOMES:
The percentage of patients whose SBP is <90 mmHg within 30 minutes of the initiation of Cleviprex infusion | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Christopher K Finch, PharmD, Principal Investigator — Methodist Healthcare, University Hospital
Locations (1):
- Methodist Healthcare, University Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Background] Pollack CV, Varon J, Garrison NA, Ebrahimi R, Dunbar L, Peacock WF 4th. Clevidipine, an intravenous dihydropyridine calcium channel blocker, is safe and effective for the treatment of patients with acute severe hypertension. Ann Emerg Med. 2009 Mar;53(3):329-38. doi: 10.1016/j.annemergmed.2008.04.025. Epub 2008 Jun 5. PMID 18534716